CLINICAL TRIAL: NCT02326064
Title: Prospective Multicenter Study in Patients With a Tumor Benign Ovarian Presumed on the Use of Algorithms Such as Roma and RMI (Risk of Malignancy Index) and Tumor Markers Such as CA125 (Cancer Antigen 125) and HE4 (Human Epididymal Protein 4)
Brief Title: Prospective Multicenter Study in Patients With a Tumor Benign Ovarian Presumed on the Use of Algorithms Such as Roma and RMI and Tumor Markers Such as CA125 and HE4
Acronym: TORCH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD064-14
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Results first posted 2024-03-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Tumor; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ovarian cancer is the fifth leading cause of cancer death in women worldwide. Most of these cancers are manifested in the form of an ovarian cyst. Practitioners are faced with two main difficulties. The first is to establish an early diagnosis. The second is to differentiate a benign tumor, a malignant tumor.

To date, there is only one biological tumor marker routinely performed before an ovarian cyst, the CA-125 (cancer antigen 125). Unfortunately, many studies have been performed and show a sensitivity and specificity unsatisfactory in view of the severity of the disease.

The principal investigator therefore propose to evaluate a new tumor marker, as well as its use in algorithms to help differentiate benign from malignant tumors, and allow earlier diagnosis in cases of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients to undergo surgery for an ovarian cyst
* presumed benign ovarian tumor (according to the rules of the IOTA(International Ovarian Tumor Analysis Group) group)
* agreement to participate in the study

Exclusion Criteria:

* pregnant patient
* minor patient
* Patient under guardianship, trusteeship, or deprived of liberty
* Patient with ascites or metastases or malignant ovarian mass presumed under the rules of IOTA group.
* Patient with an adnexal torsion is suspected
* Patient unable to understand the proposed study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized for surgery for presumed benign ovarian tumor
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, PH, Study Director — CHD Vendée
Locations (4):
- France (4):
  - Centre Hospitalier de Cholet, Cholet
  - CHD Vendée, La Roche-sur-Yon
  - CHU de Nantes, Nantes
  - CH de Saint Nazaire, Saint-Nazaire

REFERENCES:
- [Background] Dochez V, Caillon H, Vaucel E, Dimet J, Winer N, Ducarme G. Biomarkers and algorithms for diagnosis of ovarian cancer: CA125, HE4, RMI and ROMA, a review. J Ovarian Res. 2019 Mar 27;12(1):28. doi: 10.1186/s13048-019-0503-7. PMID 30917847
- [Result] Dochez V, Randet M, Renaudeau C, Dimet J, Le Thuaut A, Winer N, Thubert T, Vaucel E, Caillon H, Ducarme G. Efficacy of HE4, CA125, Risk of Malignancy Index and Risk of Ovarian Malignancy Index to Detect Ovarian Cancer in Women with Presumed Benign Ovarian Tumours: A Prospective, Multicentre Trial. J Clin Med. 2019 Oct 25;8(11):1784. doi: 10.3390/jcm8111784. PMID 31699959

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women with benign ovarian tumour | Women with borderline/ malign ovarian tumour
Started | 209 | 12
Completed | 209 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women With Benign Ovarian Tumour | Women With Borderline/ Malign Ovarian Tumour | Total
Number analyzed (Participants) | 209 | 12 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (15.1) | 53.1 (16.3) | 46.5 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 12 | 221
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Marker CA125
Description: CA125 < 35U/mL. Abnormal score if CA125 > 35U/mL.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Women with benign ovarian tumour | Women with borderline/ malign ovarian tumour
Number analyzed (Participants) | 209 | 12
U/mL | 189 (90.4) | 4 (33.3)
Statistical Analysis 1: Comparison: Women with benign ovarian tumour vs Women with borderline/ malign ovarian tumour; Test type: Superiority; p < 0.001, Mac-Nemar paired Chi-2 test

2. Primary Outcome: Tumor Marker HE4
Description: HE4 < 70 pmol/L for premenopausal women or < 140 pmol/L for postmenopausal women
  Abnormal score if HE4 > 70 pmol/L for premenopausal women or > 140 pmol/L for postmenopausal women
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Women with benign ovarian tumour | Women with borderline/ malign ovarian tumour
Number analyzed (Participants) | 209 | 12
pmol/L | 191 (91.4) | 6 (50)
Statistical Analysis 1: Comparison: Women with benign ovarian tumour vs Women with borderline/ malign ovarian tumour; Test type: Superiority; p < 0.001, Mac-Nemar paired Chi-2 test

ADVERSE EVENTS:
Description: Not applicable - not required by French law Serious adverse events and other [non-serious] events were not collected and therefore not evaluated.
Arm/Group | Women with benign ovarian tumour | Women with borderline/ malign ovarian tumour
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other